CLINICAL TRIAL: NCT00879710
Title: Effect of Diabetes Mellitus on Cholesterol Absorption, Synthesis and Statin Efficacy
Brief Title: Effect of Diabetes Mellitus on Cholesterol Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Srividya Kidambi, MD, Assistant Professor, Endocrinology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO00002485
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Hypercholesterolemia
Keywords: Diabetes Mellitus; Hypercholesterolemia; Simvastatin; Ezetimibe.
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypercholesterolemia; Diabetes Mellitus | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects with type 1 diabetes mellitus, option 1 (Other): Half the subjects will start with arm (i.e. every other subject in order)
  * Simvastatin 40 mg tablet by month daily for 6 weeks,
  * 4 weeks washout period
  Half the subjects will start with arm (i.e. every other subject in order)
  * Ezetimibe 10 mg by month for 6 weeks
  * 4 weeks washout period
  * Simvastatin 40 mg tablet by month daily for 6 weeks
  Interventions: Drug: simvastatin or ezetimibe
- Subjects with type 2 diabetes mellitus option 1 (Other): Half the subjects will start with arm (i.e. every other subject in order)
  * Simvastatin 40 mg tablet by month daily for 6 weeks,
  * 4 weeks washout period
  Half the subjects will start with arm (i.e. every other subject in order)
  * Ezetimibe 10 mg by month for 6 weeks
  * 4 weeks washout period
  * Simvastatin 40 mg tablet by month daily for 6 weeks
  Interventions: Drug: simvastatin or ezetimibe
- Subjects with type 1 diabetes mellitus, option 2 (Other): Half the subjects will start with arm (i.e. every other subject in order)
  * Ezetimibe 10 mg by month for 6 weeks,
  * 4 weeks washout period
  Interventions: Drug: simvastatin or ezetimibe
- Subjects with type 2 diabetes mellitus option 2 (Other): Half the subjects will start with arm (i.e. every other subject in order) Ezetimibe 10 mg by month for 6 weeks,
  •4 weeks washout period
  Interventions: Drug: simvastatin or ezetimibe

INTERVENTIONS:
Drug: simvastatin or ezetimibe — Subjects will be started on either simvastatin or ezetimibe (we will alternate the subjects so that half the sample will initially be treated with simvastatin and half will be started on ezetimibe). The dose of Simvastatin (Merck) is 40 mg orally at nighttime for 6 weeks and the dose of ezetimibe (Schering-Plough) is 10 mg taken orally once a day. Subjects will be instructed on low-fat diet (therapeutic life style changes diet) recommended by American Heart Association by the bionutritionist.
  Other Names: Zocor or Zetia

SUMMARY:
HMG CoA reductase inhibitors (statins) are commonly used to treat high cholesterol (HC) in both type 1 and type 2 diabetes mellitus (DM). Several studies have shown benefits of statin among patients of type 2 DM, however, no such data is available for patients with type 1 DM.

It is known from studies on cholesterol metabolism using surrogate markers that patients with type 1 DM have higher cholesterol absorption compared to normals and those with type 2 DM have higher cholesterol synthesis. Since statins inhibit synthesis, patients with type 1 DM may not have a good response and may respond better to cholesterol absorption inhibitors. The purpose of this study is to determine the cholesterol lowering effects of cholesterol absorption inhibitors and cholesterol synthesis inhibitors in subjects with type 1 and type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Hypothesis:

1. Cholesterol absorption inhibitors like ezetimibe are more effective in lowering cholesterol in subjects with type 1 diabetes mellitus . The primary outcome measures are LDL cholesterol and cholesterol tracer absorption.
2. Cholesterol synthesis inhibitors like statins are more effective in lowering cholesterol in subjects with type 2 diabetes mellitus. The primary outcomes are LDL cholesterol and 24 Hour urinary mevalonic acid levels.
3. Response to statin is related to basal cholesterol synthesis rates. The primary outcomes are LDL cholesterol and 24 Hour urinary mevalonic acid levels.
4. Response to ezetimibe is related to basal absorption rates. The primary outcome measures are LDL cholesterol, phytosterol levels and cholesterol tracer absorption.

Specific Aims:

1. Measure baseline sterol absorption using plant sterol levels and and synthesis by using 24 h excretion of urinary mevalonic acid levels in type 1 and type 2 subjects
2. Measure changes in lipid parameters, cholesterol synthesis and absorption markers in type 1 and type 2 subjects before and after 6 week therapy with simvastatin and 6 week therapy with ezetimibe after a 4 week washout period
3. Start collecting blood for future genetic analysis for polymorphisms in cholesterol absorption genes

Specific Methods:

VISIT 1: Evaluation of all the subjects that are willing to participate in the study would be carried out at the GCRC until required sample size is recruited and will include the following:

1. Sign informed consent
2. Complete a health questionnaire that has a standardized format to collect basic information regarding past and current medical history
3. Physical exam that includes measurement of blood pressure, height, weight, waist and hip circumference will be performed.
4. Blood (30ml) would be drawn for baseline chemistry including creatinine, ALT, CPK, fasting lipid panel, Apo-B, Apo A1, glycated hemoglobin (HbA1c) and serum pregnancy test in women of child bearing age. Urine will be collected for urine analysis and presence of protein in the urine
5. Evaluation of inclusion/exclusion criteria Subjects fulfilling the inclusion and exclusion criteria would be recruited into the study

Following specific procedures will be followed:

At the start of the study, subjects who are already on any lipid lowering medication will be asked to stop the medications 4 weeks prior to obtaining the baseline labs. No changes will be made to their diet, exercise pattern or in treatment for the DM. This will be done by a telephone conversation.

VISIT 2 (Day 1): Subjects will report fasting to GCRC at 8 AM. Subjects will briefly meet with bionutritionist for 24 hour dietary recall and instructions to keep a food diary on day 2 and 3. Blood sample (50ml) will be collected for fasting glucose, insulin, lipid panel, Apo B, Apo A-1, CPK, Hb A1c, plasma and serum frozen for sterol analyses (by GC) and WBC separated for DNA extraction.

The subject will be asked to consume with a cholesterol tracer (Cholesterol D5). Subjects will be asked to consume the 8 ounces in entirety. They will be asked not to eat/drink anything (except water) until the lunch time. If 8 Ounces are inadequate for breakfast, subjects will be offered another 8 Oz serving of Carnation® Instant Breakfast in the same or different flavor. If the subject is lactose intolerant, Lactaid tablets will be offered to offset the effects of milk. If subjects are unable to consume milk (with or without Lactaid®) or allergic to soy bean oil, they will be ineligible to participate in the study. Subjects will be sent home with a urine jug to collect 24-hour urine on day 3.

VISIT 3 (Day 4): Subject will bring the urine jug and food diary back for analysis and that same day will have blood (20ml) collected for evaluation of tracers. Food diary will be reviewed by the bionutritionist. Urine pregnancy test will be performed in women of child bearing age. Subjects will be started on either simvastatin or ezetimibe (we will alternate the subjects so that half the sample will initially be treated with simvastatin and half will be started on ezetimibe). The dose of Simvastatin (Merck) is 40 mg orally at nighttime for 6 weeks and the dose of ezetimibe (Schering-Plough) is 10 mg taken orally once a day. Subjects will be instructed on low-fat diet (therapeutic life style changes diet) recommended by American Heart Association by the bionutritionist.

VISIT 4 (Day 46 ± 7 days): Subjects will report fasting to GCRC at 8 AM. The subject will consume Carnation® Instant Breakfast with a cholesterol tracer (Cholesterol D5). Subjects will be asked to maintain same dietary restriction as visit 2. Subjects will be sent home with a urine jug to collect 24-hour urine on day 3. Subjects will start food diary on day 47 and 48.

VISIT 5 (Day 49 ± 7 days): Subject will bring the urine jug and food diary back for analysis and that same day will have blood (40ml) collected for evaluation of tracers, lipid panel, Apo A1, Apo B 100, ALT, CPK, plasma and serum stored for sterol analyses (by GC). Same day, weight, waist and hip circumference will be measured again. Food diary will be reviewed by bionutritionist. Subjects will be asked to bring back pill bottles also for pill count. Simvastatin or ezetimibe will be stopped for 4 weeks.

VISIT 6 (Day 77 ± 7 days): Subjects will be asked to come fasting to GCRC at 8 AM. 15ml of blood will be collected to measure lipid panel, apo B100 and Apo A1, Hb A1C, and ALT levels. Urine pregnancy test will be performed in women of child bearing age. Subjects will be started on 10 mg of ezetimibe or 40 mg of simvastatin as mentioned above for next 6 weeks.

VISIT 7 (Day 119 ± 7 days): Subjects will report fasting to GCRC at 8 AM. The subject will consume a Carnation® Instant Breakfast with cholesterol tracer (Cholesterol D5). Subjects will be asked to maintain same dietary restriction as visit 2. Subjects will be sent home with a urine jug to collect 24-hour urine on day 3.

Subjects will start food diary on day 120 and 121

VISIT 8 (Day 122 ± 7 days): Subject will bring the urine jug and food diary back for analysis and that same day will have blood (40 ml) collected for evaluation of tracers, lipid panel, Apo B100, Apo A1, Hb A1c, ALT, CPK, plasma and serum stored for sterol analyses (by GC). Weight, waist and hip circumference will be measured again. Food diary will be reviewed by bionutritionist. Ezetimibe or simvastatin therapy will be stopped. Subjects will be asked to resume their usual cholesterol lowering medications.

Ending the Study:

Study will be ended when all the required participants are enrolled. We will also consider stopping the study when accumulated data suggests that risks exceed benefits of the study or if preliminary data suggests there is a clear advantage of treating a particular group with a certain agent.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 DM:
* Age > 18 years
* Subjects diagnosed with type 1 DM (diagnosed based upon history of ketoacidosis, proven insulin dependence, absent C-peptide and or positive autoantibody profile (such as anti-GAD etc.)
* Stable A1C < 8.5%
* BMI < 31
* Type 2 DM:
* Age > 18 years
* Subjects diagnosed with type II DM (diagnosed as adult onset, not-insulin dependent and not on insulin)
* Stable A1C < 8.5%
* BMI < 31

Exclusion Criteria:

* History of active, unstable cardiovascular disease (including MI, CHF, Stroke, Angina, CABG, stenting/PTCA, peripheral vascular disease, intermittent claudication)
* Pregnancy, nursing or likely to get pregnant during the course of the study (not on oral contraceptives and premenopausal)
* Chronic Kidney Disease (creatinine > 2.0)
* Liver function test abnormalities, not previously worked up (AST or ALT >4x upper limit of normal)
* Active substance abuse including alcohol
* History of severe Hypertriglyceridemia (untreated TG > 500) and on therapy
* Use of agents that interfere with cholesterol absorption (such as fiber, resins etc.) which can not be discontinued for the duration of the study
* Actively enrolled in a weight loss program or following a special diet ( e.g.: Atkins diet)
* History of malignancy <5y
* History of Rhabdomyolysis and Myopathy
* Use of on-going oral corticosteroids
* History of HIV infection
* Use of following drugs/compounds: cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, gemfibrozil, niacin, amiodarone, verapamil or large quantities of grape fruit juice (> 1 quart per day)
* Proteinuria: more than or equal to 300mg/24 hours calculated from random urine specimen.
* BMI >31
* Anyone with hypersensitivity to either one of the study medications
* Allergy to Soy bean products
* Unable to consume milk products with or without Lactaid®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srividya Kidambi, MD, Principal Investigator — Medical College of Wisconsin; Shailendra B Patel, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin /Froedtert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Ciriacks K, Coly G, Krishnaswami S, Patel SB, Kidambi S. Effects of simvastatin and ezetimibe in lowering low-density lipoprotein cholesterol in subjects with type 1 and type 2 diabetes mellitus. Metab Syndr Relat Disord. 2015 Mar;13(2):84-90. doi: 10.1089/met.2014.0114. Epub 2014 Dec 9. PMID 25490061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertising in local news papers, Craig's list, local clinics between 2007 and 2012. Subjects were initially screened over the phone by using a telephone screening criteria (n=549). And eligible subjects (n=86) were brought to Translational Research Units (previously GCRC) for a screening visit of which 57 were enrolled.
Pre-assignment Details: After screening visit, 23 patients with type 1 diabetes, and 34 patients with type 2 diabetes were enrolled.
  All the subjects were asked to stop their lipid lowering medications for 4 weeks. All the subjects who were enrolled started the study.
Groups:
- Subjects With Type 1 Diabetes mellitus_Simva_Ezet: Subjects with T1DM were ascertained based on ketosis at the time of diagnosis and/or being treated with insulin since the diagnosis.
  All subjects were interviewed by S.K. (a board certified endocrinologist) to ensure classifications of T1DM and T2DM were accurate by history and physical exam.
  This group started with simvastatin for 6 weeks followed by 4 week washout. They were then placed on 6 weeks of ezetimibe.
- Subjects With Type 2 Diabetes mellitus_Simva_Ezet: Patients with T2DM were treated only with oral sulfonylurea drugs and/or biguanides and/or thiazolidinediones. Subjects with T2DM were excluded if they were on insulin or other injectable agents. All subjects were interviewed by S.K. to ensure classifications of T1DM and T2DM were accurate by history.
  This group started with simvastatin for 6 weeks followed by 4 week washout. They were then placed on 6 weeks of ezetimibe.
- Subjects With Type 1 Diabetes mellitus_Ezet_Simva: Subjects with T1DM were ascertained based on ketosis at the time of diagnosis and/or being treated with insulin since the diagnosis.
  All subjects were interviewed by S.K. (a board certified endocrinologist) to ensure classifications of T1DM and T2DM were accurate by history and physical exam.
  This group started with ezetimibe for 6 weeks followed by 4 week washout. They were then placed on 6 weeks of simvastatin.
- Subjects With Type 2 Diabetes mellitus_Ezet_Simva: Patients with T2DM were treated only with oral sulfonylurea drugs and/or biguanides and/or thiazolidinediones. Subjects with T2DM were excluded if they were on insulin or other injectable agents. All subjects were interviewed by S.K. to ensure classifications of T1DM and T2DM were accurate by history.
  This group started with ezetimibe for 6 weeks followed by 4 week washout. They were then placed on 6 weeks of simvastatin.
Period: Phase 1 - 6 Weeks
Arm/Group | Subjects With Type 1 Diabetes mellitus_Simva_Ezet | Subjects With Type 2 Diabetes mellitus_Simva_Ezet | Subjects With Type 1 Diabetes mellitus_Ezet_Simva | Subjects With Type 2 Diabetes mellitus_Ezet_Simva
Started | 12 (Started with simvastatin 40 mg as the starting drug) | 17 (Started with simvastatin 40 mg as the starting drug) | 11 (Started with ezetimibe 10 mg as the starting drug) | 17 (Started with ezetimibe 10 mg as the starting drug)
Completed | 10 | 14 | 9 | 13
Not Completed | 2 | 3 | 2 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Wash Out Period of 4 Weeks
Arm/Group | Subjects With Type 1 Diabetes mellitus_Simva_Ezet | Subjects With Type 2 Diabetes mellitus_Simva_Ezet | Subjects With Type 1 Diabetes mellitus_Ezet_Simva | Subjects With Type 2 Diabetes mellitus_Ezet_Simva
Started | 10 | 14 | 10 (The person who did not complete ezetimibe arm came back to complete simvastatin arm.) | 13
Completed | 10 | 14 | 10 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2 6 Weeks
Arm/Group | Subjects With Type 1 Diabetes mellitus_Simva_Ezet | Subjects With Type 2 Diabetes mellitus_Simva_Ezet | Subjects With Type 1 Diabetes mellitus_Ezet_Simva | Subjects With Type 2 Diabetes mellitus_Ezet_Simva
Started | 10 | 14 | 10 | 13
Completed | 10 | 14 | 10 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Type 1 Diabetes Mellitus,; Subjects With Type 2 Diabetes Mellitus: * Simvastatin 40 mg tablet by month daily for 6 weeks,
  * 4 weeks washout period
  * Ezetimibe 10 mg by month for 6 weeks
  simvastatin: Subjects will be started on eithersimvastatin or ezetimibe(we will alternate the subjects so that half the sample will initially be treated with simvastatin and half will be started on ezetimibe). The dose of Simvastatin (Merck) is 40 mg orally at nighttime for 6 weeks and the dose of ezetimibe (Schering-Plough) is 10 mg taken orally once a day. Subjects will be instructed on low-fat diet (therapeutic life style changes diet) recommended by American Heart Association by the bionutritionist.
- Total: Total of all reporting groups
Arm/Group | Subjects With Type 1 Diabetes Mellitus, | Subjects With Type 2 Diabetes Mellitus | Total
Number analyzed (Participants) | 23 | 34 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13) | 65 (10) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 23 | 34 | 57

OUTCOME MEASURES:

1. Primary Outcome: Changes in LDL Cholesterol
Description: Subjects with T1DM or T2DM were assigned to alternating therapy with simvastatin (40 mg) or ezetimibe (10 mg) for 6 weeks in a crossover design.
  The data are reported as follows.
  Subjects with type 1 diabetes mellitus:
  Simvastatin: Changes in LDL after 6-week therapy with simvastatin (irrespective of the treatment order) Ezetimibe: Changes in LDL after 6-week therapy with ezetimibe (irrespective of the treatment order)
  Subjects with type 2 diabetes mellitus:
  Simvastatin: Changes in LDL after 6-week therapy with simvastatin (irrespective of the treatment order) Ezetimibe: Changes in LDL after 6-week therapy with ezetimibe (irrespective of the treatment order)
Time Frame: 6 weeks after starting drug therapy
Population: We did not reach our target inclusion criteria, sample size calculations were based on assumptions.
  Our analyses after 3 years of data collection showed that we had adequate sample to answer the question we were asking. Study was terminated after 3 years with further lack of funds. Planned statistical analyses was conducted.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Subjects With Type 1 Diabetes Mellitus, | Subjects With Type 2 Diabetes Mellitus
Number analyzed (Participants) | 20 | 27
mmol/L
  simvastatin | -0.83 (0.24) | -1.47 (0.19)
  ezetimibe | -0.93 (0.23) | -0.32 (0.19)

2. Secondary Outcome: Changes in Cholesterol Absorption or Synthesis Rates From the Baseline
Description: Our plan was to measure changes in cholesterol absorption and synthesis rates from the baseline after 6 weeks of statin or ezetimibe therapy.
Time Frame: 6 weeks after initiation of drug therapy
Population: Secondary analyses were not conducted in any subjects. This is due to lack of funds.
Groups:
- Subjects With Type 1 Diabetes Mellitus; Subjects With Type 2 Diabetes Mellitus: * Simvastatin 40 mg tablet by month daily for 6 weeks,
  * 4 weeks washout period
  * Ezetimibe 10 mg by month for 6 weeks
  simvastatin: Subjects will be started on either simvastatin or ezetimibe(we will alternate the subjects so that half the sample will initially be treated with simvastatin and half will be started on ezetimibe). The dose of Simvastatin (Merck) is 40 mg orally at nighttime for 6 weeks and the dose of ezetimibe (Schering-Plough) is 10 mg taken orally once a day. Subjects will be instructed on low-fat diet (therapeutic life style changes diet) recommended by American Heart Association by the bionutritionist.
Arm/Group | Subjects With Type 1 Diabetes Mellitus | Subjects With Type 2 Diabetes Mellitus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 16 weeks (time during which participants were in the study).
Description: 16 weeks
  6 weeks of simvastatin or ezetimibe 4 weeks washout 6 weeks of simvastatin or ezetimibe
Groups:
- Subjects With Type 1 Diabetes Mellitus; Subjects With Type 2 Diabetes Mellitus: * Simvastatin 40 mg tablet/ezetimibe 10 mg by mouth daily for 6 weeks,
  * 4 weeks washout period in between
  Subjects will be started on either simvastatin or ezetimibe(we will alternate the subjects so that half the sample will initially be treated with simvastatin and half will be started on ezetimibe). The dose of Simvastatin (Merck) is 40 mg orally at nighttime for 6 weeks and the dose of ezetimibe (Schering-Plough) is 10 mg taken orally once a day. Subjects will be instructed on low-fat diet (therapeutic life style changes diet) recommended by American Heart Association by the bionutritionist.
Arm/Group | Subjects With Type 1 Diabetes Mellitus | Subjects With Type 2 Diabetes Mellitus
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/27
Other Adverse Events (participants affected / at risk) | 1/20 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Type 1 Diabetes Mellitus (N=20) | Subjects With Type 2 Diabetes Mellitus (N=27)
Intense sweating and dizziness lasting 1 hour with ezetimibe (General disorders) | 1 (1) | 0 (0) — Only one subject experienced intense sweating and dizziness lasting 1 hr with ezetimibe, and the medication was discontinued. This subject later completed the statin portion of the study.

LIMITATIONS AND CAVEATS:
1. Smaller than desirable sample size due to difficulty in recruitment.
2. Could not evaluate the effect of duration of the diabetes mellitus as independent confirmation of the duration could not be done.
3. Apolipoprotein levels were not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No